CLINICAL TRIAL: NCT05702463
Title: Assessing Pharmacokinetics and Pharmacodynamics of Daily Enteric-coated Aspirin in Patients With StablE Diabetes II
Acronym: APPEASEDII
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ICM 2023-3231
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Platelet Aggregation; Type 2 Diabetes; Aspirin; Diabetes Mellitus, Type 2; Platelet Aggregation Inhibitors
Keywords: diabetes; aspirin; Acetylsalicylic acid; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Aspirin; Mastication

STUDY DESIGN:
Intervention Model Description: triple crossover
Masking Description: laboratory personnel doing the platelet function assay will be blinded to minimize potential assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EC ASA 162 mg once daily for 7 days (Experimental): EC ASA 162 mg once daily for 7 days
  Interventions: Drug: Aspirin 162 mg EC Tab once daily for 7 days
- EC ASA 81 mg twice daily for 7 days (Experimental): EC ASA 81 mg twice daily for 7 days
  Interventions: Drug: Aspirin 81Mg Ec Tab twice daily for 7 days
- chewable ASA 40 mg twice daily for 7 days (Experimental): chewable ASA 40 mg twice daily for 7 days
  Interventions: Drug: Aspirin 40Mg Chew Tab twice daily for 7 days

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab twice daily for 7 days — Participants with incomplete platelet aggregation will be instructed to take EC ASA 81 mg twice daily for 7 days.
  Other Names: ASA 81 mg EC Tab
  Arms: EC ASA 81 mg twice daily for 7 days
Drug: Aspirin 40Mg Chew Tab twice daily for 7 days — Participants with incomplete platelet aggregation will be instructed to take chewable ASA 40 mg twice daily for 7 days.
  Other Names: ASA 40 mg Chew Tab
  Arms: chewable ASA 40 mg twice daily for 7 days
Drug: Aspirin 162 mg EC Tab once daily for 7 days — Participants with incomplete platelet aggregation will be instructed to take EC ASA 162 mg once daily for 7 days.
  Other Names: ASA 162 mg EC Tab
  Arms: EC ASA 162 mg once daily for 7 days

SUMMARY:
This phase 2 study will include patients suffering from type 2 diabetes mellitus and will first study their response to enteric coated aspirin at a dose of 80 mg per day for a 7-day period. Participants with an incomplete platelet inhibition after exposure to EC aspirin at doses of 80 mg once daily will be randomized to a random order of 3 different ASA regimens: EC ASA 162 mg once daily, EC ASA 81 mg twice daily and chewable ASA 40 mg twice daily. The aims are to determine the feasibility of a larger scale trial, and to determine the regimen associated with the lowest proportion of non-responders after randomization. Platelet function will be assessed at baseline and at day 7 of each arms of the study.

DETAILED DESCRIPTION:
APPEASED II is a triple crossover, open-label, randomized controlled pilot trial preceded by a 7-day run in period, aiming to determine the feasibility of a larger confirmatory randomized trial, and to determine the regimen associated with the lowest proportion of non-responders after randomization of EC ASA 162 mg once daily, EC ASA 81 mg twice daily and chewable ASA 40 mg twice daily in patients with type 2 diabetes.The primary endpoint will be to determine, among initial ASA non-responder participants in the run-in phase, the proportion of participants that remain ASA non-responders with different formulations and dosing regimens of ASA, including EC ASA 162 mg once daily, EC ASA 81 mg twice daily and chewable ASA 40 mg twice daily. The incomplete platelet aggregation will be evaluated by the response to arachidonic acid at a concentration of 1mM, measured by LTA (Light Transmission Aggregometry). For every platelet function assessment, serum salicylate concentration will also be measured. Upon the screening visit (day 0), blood will be drawn and baseline platelet function will be assessed. A 7 day supply of aspirin will be given to participants meeting the eligibility criteria. Participants will be instructed to take 1 dose of 80 mg of enteric coated aspirin per day at the same time every day. Upon day 7, participants will return for a second visit before the intake of their daily aspirin, and therefore 24 hours after the previous dose of aspirin was taken. Blood will be drawn and platelet function will be assessed in the same manner as described previously. Participants will then take their 7th dose of aspirin under supervision, and a blood sample will be collected and platelet function will be assessed two hours later. If participants have an incomplete platelet inhibition after exposure to EC aspirin at doses of 80 mg once daily, they will be randomized to a random order of 3 different ASA regimens: EC ASA 162 mg once daily, EC ASA 81 mg twice daily and chewable ASA 40 mg twice daily. These participants will receive the pillbox containing the first assigned regimen on this visit. The 3 study arms and the run-in phase will last 7 days each, with at least 7 days of wash-out between each arm. To accommodate participants with busy schedules and to minimize follow-up losses, a longer washout period will be tolerated if the participant is unable to return to the research center after 14 days. At every visit of the randomized portion of the trial, participants will leave with the next 6-day ASA regimen in a pillbox, that is 6 doses for the once daily regimen and 13 doses for the twice daily regimens. On day 7 of all three study arms, patients will be questioned about medication adherence with the presence of the participant's pillbox. Two blood samples will be collected, one 24 hours after the last dose and one 2 hours after taking the last dose in front of the investigators. The platelet aggregation inhibition with arachidonic acid and platelet reactivity to various agonists will be assessed by LTA. Serum levels of TxB2 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Participant must be naïve to ASA, defined as absence of chronic treatment with ASA within the previous 3 months, and of any ASA use within the previous 2 weeks;
3. Type 2 diabetes, based on at least one of the following criteria: (5)

   * Chronic treatment with oral antihyperglycemic agents or insulin therapy;
   * Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) (fasting is defined as no caloric intake for at least 8h);
   * 2-h Plasma Glucose (2h-PG) ≥ 200 mg/dL (11.1 mmol/L) during the oral glucose tolerance test (OGTT);
   * A1C ≥ 6.5% (48 mmol/ml);
4. Willing to attend all study visits of both the run-in and randomized phases of the trial.

Exclusion Criteria:

1. Definitive indication for ASA, including any evidence of clinical atherosclerotic disease, previous or current;
2. Known hypersensitivity to ASA;
3. Patient requiring dialysis;
4. Severe hepatic insufficiency or ALT > 3 x ULN;
5. High-risk GI bleeding features, such as known H. pylori infection, past or present ulcer, history of bleeding from the GI tract;
6. Bleeding diathesis;
7. Platelet count or hemoglobin levels outside of the normal reference range;
8. Planned major surgical procedure or dental procedure during the course of the study;
9. Chronic inflammatory disease requiring regular anti-inflammatory treatment;
10. Chronic treatment with an oral anticoagulant, an antiplatelet agent, NSAIDs or systemic steroids;
11. Active cancer;
12. History of hematological malignancy or myelodysplasia;
13. Pregnant or lactating women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Describe the screening rate to evaluate the feasibility of a larger scale randomized controlled trial. | 1 year
  Determine the average number of potential participants referred to us from the Montreal Clinical Research Institute (IRCM), Centre Épic, Montreal Heart Institute and the COLCOT-T2D study who are screened per month.
  Hypothesis : at least 40 potential participants per month will be screened on average
Describe the enrollment rate by the proportion of referred participants who are eligible to evaluate the feasibility of a larger scale randomized controlled trial. | 1 year
  Hypothesis : at least 70 percent of referred patients will be eligible
Describe the enrollment rate by the proportion of eligible participants who consent to evaluate the feasibility of a larger scale randomized controlled trial. | 1 year
  Hypothesis : At least 40 percent of eligible patients will give their consent to participate in the run-in phase and the study
Describe the retention rate to evaluate the feasibility of a larger scale randomized controlled trial. | 1 year
  Determine the retention rate of randomized participants
  Hypothesis : at least 85 percent of all randomized subjects will complete all study visits
Among initial ASA non-responder participants, define the proportion of participants that remain ASA non-responders with different formulations and dosing regimens of ASA. | 1 year
  Hypothesis : in at least one of the regimens studied, the proportion of ASA non-responders will be less than 50 percent.

SECONDARY OUTCOMES:
Adherence rate to study protocol | 1 year
  Hypothesis : At least 90 percent of participants will be adherent to all study doses.
Average time per participant required to complete study enrolment and all data collection. | 1 year
  Endpoints :
  Average time required to screen for, consent and enroll per participant and average time to complete study procedures and data collection per participant
Proportion of non-responders participants at day 7 of 40 mg twice daily chewable ASA regimen, 81 mg twice daily EC ASA regimen and 162 mg once daily EC ASA regimen. | 1 year
  Hypothesis: The 40 mg twice daily chewable ASA regimen will be associated with the lowest proportion of non-responders.
For the run-in phase, characterize the prevalence of ASA non-responders at steady state following a 7-day treatment with ASA EC 81 mg once daily in participants with type 2 diabetes. | 1 year
  Hypothesis: at least 10-15 percent of participants will be non-responders after taking EC ASA 81 mg die for 7 days.
Proportion of participants who are non-responders to ASA with each dose as measured by serum levels of thromboxane B2 (TxB2). | 1 year
  Non-resposne to ASA as measured by serum levels of thromboxane B2 (TxB2).
Platelet response levels to various agonists not directly related to the pharmacological target of ASA, including ADP, collagen, epinephrine and thrombin receptor-activating peptide (TRAP). | 1 year
  Non-response to ASA as measured with ADP, collagen, epinephrine and thrombin receptor-activating peptide (TRAP).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Marquis Gravel, MD, MSc, Principal Investigator — ICM Co. Ltd.
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquis-Gravel G, Roe MT, Harrington RA, Munoz D, Hernandez AF, Jones WS. Revisiting the Role of Aspirin for the Primary Prevention of Cardiovascular Disease. Circulation. 2019 Sep 24;140(13):1115-1124. doi: 10.1161/CIRCULATIONAHA.119.040205. Epub 2019 Sep 23. PMID 31545683
- [Background] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of Aspirin for Primary Prevention in Persons with Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1529-1539. doi: 10.1056/NEJMoa1804988. Epub 2018 Aug 26. PMID 30146931
- [Background] Lordkipanidze M, Pharand C, Schampaert E, Palisaitis DA, Diodati JG. Heterogeneity in platelet cyclooxygenase inhibition by aspirin in coronary artery disease. Int J Cardiol. 2011 Jul 1;150(1):39-44. doi: 10.1016/j.ijcard.2010.02.025. Epub 2010 Mar 7. PMID 20207433
- [Background] Bhatt DL, Grosser T, Dong JF, Logan D, Jeske W, Angiolillo DJ, Frelinger AL 3rd, Lei L, Liang J, Moore JE, Cryer B, Marathi U. Enteric Coating and Aspirin Nonresponsiveness in Patients With Type 2 Diabetes Mellitus. J Am Coll Cardiol. 2017 Feb 14;69(6):603-612. doi: 10.1016/j.jacc.2016.11.050. Epub 2017 Jan 11. PMID 28089180